CLINICAL TRIAL: NCT01835275
Title: Audio-enhanced Analgesia in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Randy L. Gollub, Associate Professor, MD PhD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2012P000969
Record Dates: First submitted 2013-03-29; First posted 2013-04-18 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-03

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Music conditioning (Experimental): Subjects are tested with music, sound, and silence, after conditioning to enhance music induced analgesia
  Interventions: Behavioral: Enhanced Audio; Behavioral: Audio
- Sound (Active Comparator): Subjects are tested with music, sound, and silence, after conditioning to enhance sound induced analgesia
  Interventions: Behavioral: Enhanced Audio; Behavioral: Audio
- Calibration (No Intervention): Subjects are tested with music, sound, and silence, with no enhanced audio received

INTERVENTIONS:
Behavioral: Enhanced Audio
  Arms: Music conditioning; Sound
Behavioral: Audio
  Arms: Music conditioning; Sound

SUMMARY:
The purpose of this study is to determine whether enhanced audio methods can be used to improve analgesia for experimental pain in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* 18-50 years old
* Healthy

Exclusion Criteria:

* Current diagnoses of psychiatric or neurological disorders or chronic pain
* BDI-II score greater than 13
* current or previous ear/nose/throat or hearing issues
* prior participation in pain studies
* previous advanced music training

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2012-06; Primary Completion 2013-01 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Pain Intensity and Unpleasantness | 1.5 hour testing session
  0-100 Visual Analog Scales to rate subjective pain intensity and unpleasentness

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, Mass General Hospital, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hsieh C, Kong J, Kirsch I, Edwards RR, Jensen KB, Kaptchuk TJ, Gollub RL. Well-loved music robustly relieves pain: a randomized, controlled trial. PLoS One. 2014 Sep 11;9(9):e107390. doi: 10.1371/journal.pone.0107390. eCollection 2014. PMID 25211164